CLINICAL TRIAL: NCT05606094
Title: A Multinational, Multicenter, Non-Interventional, Retrospective, Observational, Real-World Study: Treatment Patterns in Patients With HER2-Positive Locally Advanced or Metastatic Gastric or Gastroesophageal Junction Adenocarcinoma in East Asia (HER2+ GASTA Study)
Brief Title: Real-World Observational Study to Describe Treatment Patterns in Patients With HER2-Positive Locally Advanced or Metastatic Gastric or Gastroesophageal Junction Cancer in East Asia
Status: Completed | Type: Observational
Sponsor: Daiichi Sankyo Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Daiichi Sankyo (Industry)
Other Study IDs: DS-ASCAHQ-ENH-GC001
Record Dates: First submitted 2022-10-18; First posted 2022-11-04 (Actual); Last update posted 2023-12-15 (Actual); Status verified 2023-12

CONDITIONS: Gastric Cancer
Keywords: Gastric Cancer; Adenocarcinoma; Gastroesophageal Junction Adenocarcinoma
MeSH Terms: conditions — Stomach Neoplasms; Adenocarcinoma

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study will be conducted to understand real-world treatment patterns, participant characteristics (demographic and clinico-pathological characteristics), clinical outcomes and safety of different treatment regimens, and healthcare resource utilization in East Asia for HER2-positive locally advanced or metastatic gastric or gastroesophageal adenocarcinoma (de novo advanced disease, relapsed/progressed) in a real-world setting.

ELIGIBILITY:
Inclusion Criteria:

* Adult participants at the time of 1st LOT (Index Date 1e) initiation - Adult patients ≥18 years old. (Please follow local regulatory requirements if the legal age of consent for study participation is >18 years old.)
* Participants or next of kin/legal representatives who are willing to provide written informed consent as per the local regulations (if IRB/IEC/EC grants a permission to waive informed consent, it is not necessary).
* Participants who were pathologically and/or clinically diagnosed with locally advanced or metastatic gastric or gastroesophageal adenocarcinoma (de novo advanced disease, relapsed/progressed) since January 1, 2016, and its record is available at the study participating site.
* Participants whose HER2 status were pathologically confirmed HER2-positive (IHC3+ or IHC2+/ISH-positive) before/at the Index Date 2f based on the most recent archived tumor tissue sample to the Date of Diagnosisg, and its record is available at the study participating site.
* Participants who received at least 1 LOT for HER2-positive locally advanced or mGC/GEJC in an advanced setting, and its record is available at study participating site. Trastuzumab or its biosimilar use is not required.

  °Progression on or within 6 months post neoadjuvant or adjuvant therapy is counted as "rapid progressor" in a neo-adjuvant/adjuvant setting, and thus equivalent to advanced/metastatic disease failing 1 LOT.
* Participants who have at least 6 months of follow-up data from the date of 2nd LOT initiation (Index Date 2f) unless participant died within the first 6 months from the Index Date 2, and its record is available at the study participating site.

  * For rapid progressor participants in a neo-adjuvant/adjuvant setting, "Index Date 1" will be the date of neo-adjuvant treatment initiation or adjuvant treatment initiation.

Exclusion Criteria:

* Participants with a change in HER2 status from positive to negative at progression from early-stage to advanced-stage disease (change from HER2-positive to HER2-negative on repeat biopsy during treatment for advanced stage can be participated). However, if HER2-positive was confirmed before the Date of Diagnosis (or if HER2-positive was confirmed using an archived tumor tissue sample collected during early stage) and the result was followed to make the decision for the 1st LOT, this is not the case.
* Participants who had multiple cancer within 3 years of 1st LOT initiation (Index Date 1), except adequately resected melanoma skin cancer, curatively treated in-situ disease, other solid tumors curatively treated.
* Participants who are participating or have participated in an interventional study that remains blinded at time of informed consent (IC) or at the time of data collection for participants whose IC is waived by the local IRB/EC/IEC.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The target population for data collection of this study is the participants who were diagnosed with HER2-positive locally advanced or mGC/GEJC (adenocarcinoma, de novo advanced disease, relapsed/progressed), since 1 January, 2016, having completed at least 1 LOT with availability of 6 months follow-up data from the date of 2nd LOT initiation unless participant died within the first 6 months since the 2nd LOT initiation in an advanced setting in East Asia.
Sampling Method: Non-Probability Sample
Enrollment: 450 (Actual)
Dates: Start 2023-03-09 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants Receiving Each Regimen in Each Line of Treatment (LOT) | From the date of 1st line of treatment initiation to the end of follow-up, approximately 12 months
  Percentage of participants receiving each regimen in each line of treatment (LOT) since 1st LOT initiation will be assessed. LOT is defined as one regimen, possibly a combination of several drugs, given from the date of initiation of each LOT until the treatment failed to control the disease, is not tolerated by the participant, at the time of disease relapse/progression or death.
Duration of Therapy for Each Regimen | From the date of 1st line of treatment initiation to the end of follow-up, approximately 12 months
  Duration of Therapy (DoT) is defined as the length of time from initiation of each LOT to permanent discontinuation of the treatment.
Reasons for Stopping Treatments in Each Line of Treatment (LOT) | From the date of 1st line of treatment initiation to the end of follow-up, approximately 12 months
  Reasons for stopping treatments will be ascertained by patient charts and assessed by frequency and percentage.
Treatment Sequencing Pathways | From the date of 1st line of treatment initiation to the end of follow-up, approximately 12 months
  Treatment sequencing from 1st LOT to 2nd LOT and to the subsequent LOT will be assessed.
Percentage of Participants Receiving Locoregional Treatment for Localized Disease and Metastasis (Radiotherapy and/or Surgery) | From the date of 1st line of treatment initiation to the end of follow-up, approximately 12 months
  Percentage of participants receiving locoregional treatment for localized disease and locoregional treatment for metastasis (radiotherapy and/or surgery) since 1st LOT initiation will be assessed.

SECONDARY OUTCOMES:
Real World Progression Free Survival | From the date of 1st line of treatment initiation to the end of follow-up, approximately 12 months
  Length of time from the date of initiation of LOT to the date of real-world disease progression or death due to any cause, whichever comes first.
Real Word Overall Survival | From the date of 1st line of treatment initiation to the end of follow-up, approximately 12 months
  Length of time from the date of initiation of LOT to death due to any cause.
Real World Time to Treatment Failure | From the date of 1st line of treatment initiation to the end of follow-up, approximately 12 months
  Length of time from the initiation of LOT to the date of real-world disease progression, treatment discontinuation, or death due to any cause, whichever occurs first.
Real World Time to Discontinuation | From the date of 1st line of treatment initiation to the end of follow-up, approximately 12 months
  Length of time from the date the participant initiates the LOT to the date the participant discontinues that LOT or death due to any cause, whichever occurs first.
Real-world Time to Next Treatment | From the date of 1st line of treatment initiation to the end of follow-up, approximately 12 months
  Length of time from the date the participant initiates the LOT to the date the participant initiates next LOT or death from any cause, whichever occurs first.
Real Word Objective Response Rate | From the date of 1st line of treatment initiation to the end of follow-up, approximately 12 months
  Proportion of participants who achieved real-world complete response or real-world partial response to treatment for each LOT.
Real World Disease Control Rate | From the date of 1st line of treatment initiation to the end of follow-up, approximately 12 months
  Proportion of participants with real-world complete response, real-world partial response and real-world stable disease during treatment for each LOT.
Number of Deaths in Each Line of Treatment | From the date of 1st line of treatment initiation to the end of follow-up, approximately 12 months
Cause of Death in Each Line of Treatment | From the date of 1st line of treatment initiation to the end of follow-up, approximately 12 months
Number of Participants with Adverse Events of Special Interest (AESI) In Each Line of Treatment | From the date of 1st line of treatment initiation to the end of follow-up, approximately 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Study Leader, Study Director — Daiichi Sankyo
Locations (31):
- China (8):
  - Sichuan Cancer Hospital, Chengdu
  - Sun Yat-sen University Cancer Center, Guangdong
  - The First Affiliated Hospital of Anhui Medical University, Hefei
  - Hubei Cancer Hospital, Hubei
  - Shanghai Changhai Hospital, Shanghai
  - Tianjin Medical University Hospital, Tianjin
  - Second Affiliated Hospital ZheJiang University School of Medicine, Zhejiang
  - Henan Cancer Hospital, Zhengzhou
- Hong Kong (3):
  - Queen Mary Hospital, Pok Fu Lam
  - Prince of Wales Hospital, Shatin
  - Tuen Mun Hospital, Tuenmen
- South Korea (10):
  - Dong-A University Hospital, Busan
  - Chungbuk National University Hospital, Cheongju-si
  - Kyungpook National University Chillgok Hospital, Deagu
  - Pusan National University Yangsan Hospital, Gyeongsangnam-do
  - Kangbuk Samsung Hospital, Seoul
  - Samsung Medical Center, Seoul
  - Chung-Ang University Hospital, Seoul
  - Korea University Anam Hospital, Seoul
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Seoul
- Taiwan (10):
  - Chiayi Chang Gung Memorial Hospital, Chiayi City
  - Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City
  - Kaohsiung Medical University Hospital, Kaohsiung City
  - China Medical University Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - Chi Mei Medical Center, Tainan
  - Taipei Veterans General Hospital, Taipei
  - Koo Foundation Sun Yat-Sen Cancer Center, Taipei
  - MacKay Memorial Hospital, Taipei
  - Linkou Chang Gung Memorial Hospital, Taoyuan District

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) on completed studies and applicable supporting clinical trial documents may be available upon request at https://vivli.org/. In cases where clinical trial data and supporting documents are provided pursuant to our company policies and procedures, Daiichi Sankyo will continue to protect the privacy of our clinical trial participants. Details on data sharing criteria and the procedure for requesting access can be found at this web address: https://vivli.org/ourmember/daiichi-sankyo/
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Completed studies that has reached a global end or completion with all data set collected and analyzed, and for which the medicine and indication have received European Union (EU) and United States (US), and/or Japan (JP) marketing approval on or after 01 January 2014 or by the US or EU or JP Health Authorities when regulatory submissions in all regions are not planned and after the primary study results have been accepted for publication.
Access Criteria: Formal request from qualified scientific and medical researchers on IPD and clinical study documents on completed clinical trials supporting products submitted and licensed in the United States, the European Union and/or Japan from 01 January 2014 and beyond for the purpose of conducting legitimate research. This must be consistent with the principle of safeguarding study participants' privacy and consistent with provision of informed consent.
URL: https://vivli.org/ourmember/daiichi-sankyo/